CLINICAL TRIAL: NCT00250887
Title: A Phase II Open Label Study of the Pre- and Postoperative Use of ZD1839 (Iressa) in Recurrent Glioblastoma, Including Translational Research
Brief Title: Pre- and Postoperative Use of ZD1839 (Iressa) in Recurrent Glioblastoma, Including Translational Research
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0526
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2007-10

CONDITIONS: Recurrent Glioblastoma
Keywords: recurrent Glioblastoma, Gefitinib
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gefitnib

SUMMARY:
This study aims to determine effectiveness of Gefitinib (Iressa) in recurrent glioblastoma after standard treatment (surgery, radiationtherapy and at least a first line chemotherapy). Gefitinib is a specific inhibitor of the epidermal growth factor receptor (EGFR). EGFR is elevated in more than 50% of malignant gliomas. At recurrence, secondary surgery and pre- and postoperative Gefitinib is offered to patients in good performance status. Clinical outcome of patients and correlation to translational research will be evaluated.

DETAILED DESCRIPTION:
Glioblastoma (GBM) patients who relapse and are in good performance status, without serious neurological deficits are offered secondary surgery and participation in the trial. Eligible patients must have had standard treatment including primary surgery, radiation therapy and at least a first line chemotherapy. Patients on cytochrome P450 isoenzyme CYP3A4-inducing antiepileptic drugs (EIAE) are excluded due to ensuing interactions of these drugs with gefitinib metabolism, reducing systemic availability. After giving written informed consent, patients receive gefitinib 500 mg daily starting at least 5 days prior to re-operation, allowing a steady state condition.Treatment continues until tumor progression or occurrence of intolerable side effects.The specimens collected at surgery will undergo translational research, aiming to correlate drug accumulation and molecular signatures of GBM samples with clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* recurrent glioblastoma
* informed consent
* reoperation planned
* fresh frozen sample obtainable

Exclusion Criteria:

* enzyme inducing antiepileptic drugs
* pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-07; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
molecular signature of EGFR responsiveness to ZD1839

SECONDARY OUTCOMES:
PFS

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Hofer, MD, Principal Investigator — University Hospital, Zürich
Locations (1):
- University Hospital Zürich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Hegi ME, Diserens AC, Bady P, Kamoshima Y, Kouwenhoven MC, Delorenzi M, Lambiv WL, Hamou MF, Matter MS, Koch A, Heppner FL, Yonekawa Y, Merlo A, Frei K, Mariani L, Hofer S. Pathway analysis of glioblastoma tissue after preoperative treatment with the EGFR tyrosine kinase inhibitor gefitinib--a phase II trial. Mol Cancer Ther. 2011 Jun;10(6):1102-12. doi: 10.1158/1535-7163.MCT-11-0048. Epub 2011 Apr 6. PMID 21471286